CLINICAL TRIAL: NCT00923182
Title: A Japanese Phase I Study of Alemtuzumab in Japanese Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: A Safety Confirmatory Study of Alemtuzumab in Japanese Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMCLL07709; 14020
Record Dates: First submitted 2009-06-09; First posted 2009-06-18 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: Relapsed or Refractory Chronic Lymphocytic Leukemia,; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab (Experimental): The starting dose of alemtuzumab was 3 mg. The dose was gradually escalated on a daily basis (3 mg, 10 mg, and then 30 mg) until the patient tolerated a dose of 30 mg IV infusion over 2 hours. All subsequent doses of alemtuzumab were 30 mg IV 3 times a week (every other day).
  Interventions: Drug: alemtuzumab

INTERVENTIONS:
Drug: alemtuzumab
  Other Names: MabCampath, BAY86-5045, CAMPATH-1H

SUMMARY:
The primary objective of this study is to confirm the safety profile of alemtuzumab 30 mg (the US/European Union (EU) approved dose) in Japanese patients with relapsed or refractory Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
NOTE: This study was previously posted by Bayer. In December 2009, this study was acquired by Genzyme Corporation. Genzyme Japan K.K. is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* B-cell Chronic Lymphocytic Leukemia (B-CLL) according to the 1996 National Cancer Institute-sponsored Working Group (NCI-WG) Criteria
* One or more, but <= 3 previous treatment regimens for Chronic Lymphocytic Leukemia (CLL)
* Patient requires treatment for CLL (Rai stage III and IV disease or stage 0 to II disease with evidence of progression)
* Adequate bone marrow, liver and renal function
* More than 4 weeks since prior chemotherapy or chemoimmunotherapy, including investigational agents, for the treatment of CLL. Patient must have recovered from the acute side effects incurred as a result of previous therapy
* World Health Organization (WHO) Performance Status (PS) 0,1
* Life expectancy of at least 24 weeks
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 2 weeks after the completion of trial
* Written informed consent

Exclusion Criteria:

* Known human immunodeficiency virus (HIV) seropositivity
* Active hepatitis or a history of prior viral hepatitis B or hepatitis C, or positive hepatitis B serologies. Patients with a positive hepatitis B surface antibody (HBsAb) test with a documented history of prior hepatitis B immunization are eligible as long as other criteria are met (i.e., negative tests for : hepatitis B surface antigen [HBsAg], hepatitis B core antibody [HBcAb] and hepatitis C virus antibody [HCVAb])
* Active uncontrolled infection
* Recent documented history (within 2 years) of active tuberculosis (TB), current active TB infection, currently receiving anti-tuberculous medication (e.g., isoniazid, rifampin, streptomycin, pyrazinamide, or others)
* Positive cytomegalovirus (CMV) by Polymerase Chain Reaction (PCR) assay
* Transformation to aggressive lymphoma (e.g., Richter's syndrome)
* Past history of anaphylaxis following exposure to humanized monoclonal antibodies
* Previous treatment with alemtuzumab
* Previous hematopoietic stem cell transplant
* Pregnant or breast-feeding patients
* Central nervous system (CNS) involvement with CLL
* Other severe, concurrent diseases (e.g., cardiac or pulmonary disease), mental disorders, or major organ malfunction (e.g., liver, kidney) that could interfere with the patient's ability to participate in the study
* Medical condition requiring chronic use of oral corticosteroids at a dose higher than physiologic replacement.
* Active malignancy, other than CLL, which needs therapy with anti-cancer drug(s)
* Autoimmune anemia and/or thrombocytopenia
* Small lymphocytic lymphoma

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety profile: As measured by physical examinations, vital signs, adverse events, concomitant medications and laboratory tests | Until 24 weeks after end of treatment

SECONDARY OUTCOMES:
Overall response rate: Defined as the proportion of patients who achieved complete remission (CR) or partial remission (PR) as the best response according to the investigator's determination using the NCIWG response criteria | Until 24 weeks after end of treatment
Pharmacokinetic profiles: Area under the serum concentration vs time curve over the dosing interval, Maximum drug concentration in serum, terminal elimination half-life following the last dose, total body clearance and volume of distribution | until 24 weeks after end of treatment
Time to response: Defined as the time from date of initial treatment until first objective documentation of response (CR or PR) as determined by the investigator. | Until 24 weeks after end of treatment
  If a patient achieves PR before CR, the onset date of PR will be used in the calculation
Duration of response: Defined as the time from first objective documentation of response (CR or PR) by the investigator to first objective documentation of progressive disease by the investigator | Until 24 weeks after end of treatment
Time to progression: Defined as the time from date of initial treatment to first objective documentation of progressive disease by the investigator | Until 24 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- Japan (6):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Tsukuba, Ibaraki
  - Sendai, Miyagi
  - Bunkyo-ku, Tokyo
  - Chuo-ku, Tokyo

REFERENCES:
- [Derived] Ishizawa K, Fukuhara N, Nakaseko C, Chiba S, Ogura M, Okamoto A, Sunaga Y, Tobinai K. Safety, efficacy and pharmacokinetics of humanized anti-CD52 monoclonal antibody alemtuzumab in Japanese patients with relapsed or refractory B-cell chronic lymphocytic leukemia. Jpn J Clin Oncol. 2017 Jan;47(1):54-60. doi: 10.1093/jjco/hyw146. Epub 2016 Oct 7. PMID 28122892